CLINICAL TRIAL: NCT00954057
Title: A Single-masked, Placebo Controlled, Multi-center Pilot Study to Determine the Safety and Efficacy of Orbital Injections of a Fixed Dose of LIPO-102 in Patients With Symptomatic Exophthalmos Associated With Thyroid-related Eye Disease
Brief Title: Pilot Study to Determine Safety and Efficacy of Orbital Injections of LIPO-102 in Patients With Symptomatic Exophthalmos Associated With Thyroid-related Eye Disease (TED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neothetics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LIPO-102-CL-06
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Thyroid-Related Eye Disease
Keywords: TED

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- LIPO-102 (Experimental): Intraorbital Injection
  Interventions: Drug: LIPO-102
- Placebo (Placebo Comparator): Intraorbital Injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LIPO-102 — intraorbital injection
  Arms: LIPO-102
Drug: Placebo — intraorbital injection
  Arms: Placebo

SUMMARY:
This is a pilot study to determine the safety and efficacy of orbital injections of LIPO-102.

ELIGIBILITY:
Inclusion Criteria:

* Male or Non pregnant female
* Symptomatic exophthalmos
* Inactive Thyroid Eye Disease
* Signed informed consent

Exclusion Criteria:

* Known hypersensitivity to study drugs
* Treatment with an investigational agent within 30 days of first dose
* History of Thyroid Eye Disease less than 6 months
* Previous decompression surgery
* Glaucoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Safety: physical examinations, laboratory tests, VISA activity score, AE assessments | 8 weeks treatment and 1 week follow up

SECONDARY OUTCOMES:
Efficacy: change in proptosis, VISA activity score, VAS for Eye Appearance Satisfaction | 8 weeks treatment and 1 week follow up

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (4):
  - Adelaide
  - Brisbane
  - Melbourne
  - Sydney
- Auckland, New Zealand